CLINICAL TRIAL: NCT03187288
Title: An Open-Label, Dose Escalation, Safety and Pharmacokinetic Study of CFI-400945 Fumarate Administered Orally to Patients With Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome
Brief Title: Study of CFI-400945 Fumarate in Patients With Relapsed or Refractory AML or MDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFI-400945-CL-002
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndromes; Relapsed Cancer; Refractory Cancer
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Recurrence; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CFI-400945 (Experimental): CFI-400945 will be given by mouth at 64,96,128,160,192 or 224 mg/day, everyday until intolerable side effects or disease progression.
  Interventions: Drug: CFI-400945 Fumarate

INTERVENTIONS:
Drug: CFI-400945 Fumarate — CFI-400945 is an investigational drug that is being look at for the treatment of acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS). CFI-400945 is an oral (taken by mouth) drug that blocks Polo-like kinase 4 (PLK4) activity. PLK4 is a protein that is important in regulating cell growth and division and cell death. Many tumors are shown to make too much PLK4. When there is too much PLK4 produced, it is believed to contribute to uncontrolled cancer cell growth and division. Therefore, by blocking this protein from working, it is believed to stop tumors from growing or shrink them.

SUMMARY:
This is a phase 1 study of investigational drug CFI-400945 in patients with relapsed or refractory acute myeloid leukemia or myelodysplastic syndrome. The purpose of this phase 1 study is to see how safe and tolerable the study drug is and to determine the best dose (maximum tolerated dose or recommended phase 2 dose) that can be given in this patient population.

DETAILED DESCRIPTION:
Participants will be screened prior to the start of the study drug for eligibility.

Eligible participants will take CFI-400945 by mouth, once a day, every day of each 28 day cycle. Participants will be asked to keep a study drug diary.

While receiving the study drug, participants will have standard tests and procedures done for safety purposes.

Procedures for research purposes include bone marrow aspirate and additional blood collection for biomarker research, and additional blood samples for pharmacokinetic research.

When participants stop the study drug permanently for any reason, they will be asked to have an End of Treatment Visit and be followed for safety purposes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Relapsed and/or refractory myeloid leukemia (AML) or myelodysplastic syndrome (MDS) that meets certain criteria for prior treatments
* Have acceptable circulating blasts count
* Have clinically acceptable laboratory blood and urine test results
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Be able to swallow oral medications
* Have a life expectancy of 3 months or more
* Agree to use highly effective means of contraception during a defined period
* Negative serum pregnancy test before the start of the study drugs
* Have the ability to understand the requirements of the study, provide written informed consent which includes authorization for release of protected health information, abide by the study restrictions, provide a blood and bone marrow sample for genetic testing and agree to return for the required assessments

Exclusion Criteria:

* Have received cancer therapies within 14 days or 5 half-lives (whichever is shorter) prior to first dose of study drug or have not recovered from toxicities from prior treatments
* Not recovered from toxicities related to allogeneic transplant
* Known active extramedullary central nervous system (CNS) AML
* Secondary cancer needing therapy with exceptions
* Known active human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection
* Known significant mental illness or other condition that may affect the ability to follow the requirements of the study
* Have a chronic infection
* Have uncontrolled severe hypertension
* Have symptomatic congestive heart failure
* Have active angina pectoris or recent myocardial infarction
* Have chronic atrial fibrillation or unacceptable QTc
* Have had major surgery within 21 days of starting therapy
* Have additional uncontrolled serious medical or psychiatric illness
* Have any medical condition that would affect taking the study drug
* Receiving treatment with full dose warfarin
* Receiving treatment with drugs not allowed in this study
* Women who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the frequency and severity of treatment-emergent adverse events in patients | 5 years
  This will be done to assess safety and tolerability of CFI-400945 fumarate
Highest tolerated dose of CFI-400945 fumarate | 5 years
  The Maximum Tolerated Dose MTD is defined as the highest dose level that does not lead to unacceptable toxicity in two or more patients in a dosing cohort.
Recommended phase 2 dose of CFI-400945 fumarate | 5 years
  Following completion of dosing of at least 1 cycle for all patients enrolled the Recommended Phase 2 Dose (RP2D) will be determined.It will be based upon the MTD established during dose escalation and its comprehensive outcome

SECONDARY OUTCOMES:
Number of participants with response to treatment | 5 years
  Patients responses will be assess using the International Working Group response criteria for AML and MDS.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yee, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (2):
- Canada (2):
  - Juravinski Hospital and Cancer Centre, Hamilton, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No